CLINICAL TRIAL: NCT04304378
Title: Enhancing Capacity for Mental Health Research and Care in Cambodia: Trauma Informed Treatment Algorithms for Novel Outcomes
Brief Title: Trauma Informed Treatment Algorithms for Novel Outcomes
Acronym: TITAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, St. Louis (Other)
Collaborators: NCHADS - Ministry of Health of Cambodia (Other); Royal University of Phnom Penh (Unknown); Florida International University (Other); Center for Trauma and Research Organization (CTRO Cambodia) (Unknown); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert Paul, Curators' Distinguished Professor, University of Missouri, St. Louis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH114722 (NIH); R01MH114722 (NIH)
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Randomized controlled trial; Post-traumatic stress disorder; Global health; Mental disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization Techniques (ST) (Active Comparator): Participants randomized into ST will receive 6 weekly 1-hour sessions of Stabilization Techniques from a Khmer-speaking mental health professional. Sessions provide an opportunity to improve emotion regulation and provide coping skills for managing symptoms of PTSD.
  Participants will complete a follow-up assessment 2 months after randomization in which PTSD symptoms will be re-assessed using the PTSD Checklist (PCL-5) for the Diagnostic and Statistical Manual for Mental Disorders (DSM-5). Those who exhibit a 50% reduction in PTSD symptoms from baseline and no longer meet criteria for PTSD will be designated as responders and will receive no further treatment. Participants who continue to display clinically meaningful elevations in PTSD symptoms (i.e., non-responders) will receive EMDR, which is the standard of care for trauma treatment in Cambodia. EMDR sessions will be delivered by a Khmer-speaking mental health professional.
  Interventions: Behavioral: Stabilization Techniques (ST); Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)
- Stabilization Techniques with Behavioral Activation (ST+BA) (Experimental): Participants randomized into ST+BA will receive 3 weekly 1-hour sessions of ST and 3 weekly 1-hour sessions of BA from a Khmer-speaking mental health professional. Sessions include stabilization techniques and behavioral skills that aim to establish and maintain routines, reduce avoidance, and manage negative emotions.
  Participants will complete a follow-up assessment 2 months after randomization in which PTSD symptoms will be re-assessed using the PTSD Checklist (PCL-5) for the Diagnostic and Statistical Manual for Mental Disorders (DSM-5). Those who exhibit a 50% reduction in PTSD symptoms from baseline and no longer meet criteria for PTSD will be designated as responders and will receive no further treatment. Participants who continue to display clinically meaningful elevations in PTSD symptoms (i.e., non-responders) will receive EMDR, which is the standard of care for trauma treatment in Cambodia. EMDR sessions will be delivered by a Khmer-speaking mental health professional.
  Interventions: Behavioral: Stabilization Techniques with Behavioral Activation (ST+BA); Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Behavioral: Stabilization Techniques (ST) — The Stabilization Techniques intervention provides an opportunity to improve emotion/affect regulation and coping skills. The overarching goal of these sessions is to introduce different ways of managing emotional distress through imagery and stress reduction techniques. ST sessions focus on providing coping mechanisms for managing important symptoms of PTSD (i.e., hyperarousal, negative emotions, and physical symptoms).
  Arms: Stabilization Techniques (ST)
Behavioral: Stabilization Techniques with Behavioral Activation (ST+BA) — The Stabilization Techniques with Behavioral Activation intervention includes stabilization techniques as well as sessions targeted at increasing time engaged in physical activities during times outside of the intervention session. Preferred activities are selected by the participant. Strategies to foster engagement in the selected activities will include self-monitoring, structuring and scheduling daily activities, rating the degree of pleasure and accomplishment experienced during engagement in specific daily activities, exploring alternative behaviors related to achieving goals, and using role-play to address specific barriers. Establishing/maintaining routines and behavioral strategies to reduce avoidance and mange negative emotions are emphasized.
  Arms: Stabilization Techniques with Behavioral Activation (ST+BA)
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — EMDR is an exposure-based treatment that is the standard of care for PTSD delivered by the research team in Phnom Penh. EMDR utilizes sensory stimulation when participants are engaged in mental processing of traumatic material. EMDR follows a sequential framework targeting 1) past memories, 2) present symptoms, and 3) future actions.

SUMMARY:
This randomized controlled trial (RCT) will examine the feasibility, acceptability, and preliminary efficacy of a beginning treatment for Post-Traumatic Stress Disorder (PTSD) with Behavioral Activation (BA). Cambodian men and women who screen positive for PTSD will be randomized to receive six individually delivered sessions of either: 1) Stabilization Techniques alone (ST); or 2) ST+BA. After two months, all participants who continue to report clinically meaningful elevations in PTSD will receive Eye Movement Desensitization Reprocessing (EMDR). All participants will complete a follow-up assessment at four months post-randomization.

DETAILED DESCRIPTION:
Nearly half of the Cambodian population reports elevated levels of psychological distress and PTSD. The high levels of psychological distress are linked directly to the report of remote and more recent trauma exposures, the most notable of which is the agrarian political regime of the Khmer Rouge during the 1970s, which occurred in the aftermath of the Vietnam War. During this period, approximately 1.5 million Cambodian residents died of starvation and sickness, 500,000 individuals were executed, and another two million were displaced over the course of several years. Political stability took shape in the early 1990s after the enactment of the United Nations Transitional Authority in Cambodia. However, the prior violence undermined an already fragile healthcare system, including mental health institutions and physicians providing direct patient care.

The combination of high trauma exposure, sustained conflict, and limited psychiatric capacity has created heightened vulnerability for Cambodians, and the need to assist those struggling with PTSD. There is a pressing need to reverse this trajectory using novel approaches to address mental health needs that are effective and scalable, providing a strong basis to conduct the proposed work in Cambodia. In partnership with the Cambodian Department of Mental Health and Substance Abuse, Ministry of Health, this NIH-sponsored study will examine the feasibility, acceptability, and preliminary efficacy integrating BA into trauma treatment that is being delivered by the Mekong Project in Cambodia.

ELIGIBILITY:
Inclusion Criteria:

* Trauma exposure and screens positive for PTSD as measured by the DSM-5 PTSD Checklist (PCL-5), a 20-item scale to measure severity of PTSD symptoms
* Able to communicate in Khmer
* Able to provide informed consent as defined by ability to accurately paraphrase the purpose

Exclusion Criteria:

* Active psychosis or developmental disorder that precludes an individual's ability to provide informed consent
* Severe alcohol or substance use disorder a determined by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST)

Note:

* Use of psychiatric medications will be allowed but our preliminary work revealed fewer than 5% of all individuals receive medications for PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Percent of study participants who no longer screen positive for PTSD at four months using the PCL-5 questionnaire. | 4 months

SECONDARY OUTCOMES:
Culturally-Relevant PTSD Symptoms | 4 months
  The Cambodian Symptom and Syndrome Inventory (CSSI) is a culturally validated measure of PTSD symptoms that yields a total score ranging from 0-148, with higher scores indicative of greater symptomatology.
Psychological Distress | 4 months
  The Depression, Anxiety and Stress Scale (DASS-21) is a validated measure of psychological distress that yields domain scores ranging from Normal (depression=0-4; anxiety=0-3; stress=0-7) to Extremely Severe (depression=14+; anxiety=10+; stress=17+).
Alcohol and Substance Use | 4 months
  The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) provides validated composite scores indexing the severity of alcohol and other substance use (Mild = 0-3; Moderate = 4-26; Severe = 27 or greater).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paul, Ph.D., Principal Investigator — University of Missouri, St. Louis
Locations (2):
- Cambodia (2):
  - Center for Trauma Care and Research Organization, Phnom Penh
  - EMDR Association Office, Phnom Penh

REFERENCES:
- [Derived] Bertram JE, Kryah R, Vandermause R, Ean N, Paul R, Carrico A, Sophal C, Bruce S, Gregory K, Stein E, Mannarino J. "No matter what, we just work with the trauma...": Mental Health Therapists' Care of Diverse Sexual and Gender Identity Citizens in Cambodia. Res Sq [Preprint]. 2023 Feb 20:rs.3.rs-2584144. doi: 10.21203/rs.3.rs-2584144/v1. PMID 36865179